CLINICAL TRIAL: NCT03925324
Title: A Randomized, Double-Blind, Placebo-Controlled Phase IIa Study of the Safety and Efficacy of Intravenous Delivery of Allogeneic Mesenchymal Stem Cells in Cardiomyopathy Patients and Implanted Left Ventricular Assist Device
Brief Title: Serial Infusions of Allogeneic Mesenchymal Stem Cells in Cardiomyopathy Patients With Left Ventricular Assist Device
Acronym: STEM-VAD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding/Covid-19
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STEMVAD-001
Record Dates: First submitted 2019-04-01; First posted 2019-04-24 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Ischemic Heart Disease; Non-ischemic Cardiomyopathy
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) (Experimental): Three intravenous infusions of 1.5 million (aMBMC) per kg administered at approximately 2mL/min. Maximum dose as for 100kg subject or 150 million cells for any subject 100kg or more with each infusion 1 month apart.
  Interventions: Biological: Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC)
- Placebo (Placebo Comparator): Three intravenous infusions of 1.5 mL/kg Lactated Ringer's Solution with each infusion 1 month apart.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) — Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) 1.5 million cells/kg
  Arms: Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC)
Other: Placebo — 1.5 mL/kg Lactated Ringer's Solution
  Arms: Placebo

SUMMARY:
A study to assess the safety and preliminary efficacy of serial intravenous dose of Allogeneic Mesenchymal Bone Marrow Cells in subjects with heart failure and implanted left ventricular assist devices.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, single-center, randomized study to assess the safety and preliminary efficacy of a three serial intravenous doses of allogeneic mesenchymal bone marrow cells to subjects with heart failure and implanted left ventricular assist devices.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Advanced Heart Failure
3. Advanced HF defined as HF requiring LVAD implantation and deemed stable on his/her LVAD.
4. On stable medical therapy (per the discretion of the treating physician) including beta-blockers, ACE-inhibitors, angiotensin receptors blockers, angiotensin receptor neprilysin inhibitor, mineralocorticoid receptor antagonists, isosorbide, hydralazine, and mineralocorticoid receptor antagonists) and optimized pump speed for at least a month prior to randomization.
5. HS-CRP level≥2 mg/l.
6. NYHA class II-III symptoms.
7. Ability to understand and provide signed informed consent.
8. Reasonable expectation that patient will receive standard post-treatment care and attend all scheduled safety follow-up visits

Exclusion Criteria:

1. Women of childbearing potential. Postmenopausal women or women with permanent contraception method (defined as total hysterectomy) will not be excluded.
2. History of debilitating stroke (modified Rankin Score > 3) within 3 months.
3. The likelihood of requirement of cardiac surgery during the study period.
4. Presence of clinically significant, uncorrected left sided valvular heart disease, active acute myocarditis, or uncontrolled hypertension defined as Persistently elevated mean arterial blood pressure (>100 mmHg). Echocardiography within 12 months of screening. Patients can be re-evaluated, at the discretion of the investigator.
5. QTc >550 ms (in the absence of bundle branch block, interventricular conduction delay or ventricular pacing). Electrocardiogram (ECG) within 60 days.
6. History of cardiac arrest within 3 months.
7. Hypertrophic or infiltrative cardiomyopathy.
8. Considered or listed for organ transplantation or history of organ transplantation
9. Illness other than HF with life expectancy less than 12 months.
10. Enrolled in an interventional trial or received an experimental drug or device within 30 days of randomization.
11. Left ventricular assist device implantation >2 years prior to enrollment.
12. Biventricular assist device (Bi-VAD) support.
13. Severe COPD defined by FEV1<1L, FEV1/FVC<70% within 12 months if known history of COPD, otherwise FEV1<1L, FEV1/FVC<70% within 24 months
14. Uncontrolled seizure disorder.
15. Clinically significant hematologic, hepatic, or renal impairment as determined by screening clinical laboratory tests within the last 30 days:

    Liver disease = ALT or AST > 3x normal, alkaline phosphatase or bilirubin >2x normal Renal disease = on long term dialysis Hematologic = Unexplained persistent leukocytosis (WBC >11 K/UL) or hemoglobin < 8.5 gm/dl
16. Presence of any other clinically-significant medical condition, psychiatric condition, or laboratory abnormality, that in the judgment of the investigator or sponsor may affect compliance with the study protocol or pose a safety risk to the subject.
17. Inability to comply with the conditions of the protocol.
18. Acute coronary syndrome within 4 weeks (clinical diagnosis, confirmed by electrocardiographic abnormalities and elevation of troponin-I).
19. Malignancy within the previous five years, except adequately treated basal cell carcinoma, provided that it is neither infiltrating nor sclerosing, and carcinoma in situ of the cervix.
20. Active uncontrolled systemic infection. Positive blood or deep tissue cultures or clinical or imaging evidence of systemic infection despite complete course of effective antimicrobial therapy as determined by infectious diseases. Localized (non-systemic) infection is not an exclusion criterion. Patients can be re-evaluated, at the discretion of the investigator.
21. Early postpartum cardiomyopathy (within six months of diagnosis).
22. Presence of inherited or acquired immune deficiency or human immunodeficiency virus infection (HIV). Negative HIV test within the preceding 12 months is required.
23. Systemic corticosteroids, immunosuppressive drug therapy (cyclophosphamide, methotrexate, cyclosporine, tacrolimus, azathioprine, mycophenolate, sirolimus, etc.), and DNA depleting or cytotoxic drugs taken within four weeks prior to study treatment.
24. Known Porphyria.
25. Allergy to sodium citrate or any caine type of local anesthetic.
26. Patient enrolled in hospice care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Temperature
Description: Temperature
Time Frame: up to 12 months post enrollment
Population: Due to study termination and small sample size, no analysis was performed
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Uncontrolled Systemic Infection
Description: Number of admission for uncontrolled systemic infection
Time Frame: up to 12 months post enrollment
Population: Due to study termination and small sample size, no analysis was performed
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: All-cause Mortality
Description: Rate of Death
Time Frame: up to 12 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
Number analyzed (Participants) | 2 | 2
Participants | 1 | 1

4. Secondary Outcome: NK Cell Depletion
Description: percent reduction in NK cells
Time Frame: Baseline to day 90
Population: Due to study termination and small sample size, no analysis was performed
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in the Following Cardiac Biomarker
Description: The change in the lab values N-Terminal Prohormone of Brain Natriuretic Peptide (NT-ProBNP)
Time Frame: Baseline and day 90 post initial infusion
Population: Due to study termination and small sample size, no analysis was performed
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in RV Systolic Function
Description: Change in RV systolic function
Time Frame: Baseline and day 90 post initial infusion
Population: Due to study termination and small sample size, no analysis was performed
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Hospitalizations Due to Right Heart Failure
Description: Number of hospitalizations for to right heart failure
Time Frame: day 90
Population: Due to study termination and small sample size, no analysis was performed
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: 6 Minute Walk Distance Changes
Description: 6 minute walk distance changes
Time Frame: Baseline and day 90 post initial infusion
Population: Test was not performed for any subjects at 90 days, therefore no changes could be analyzed
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Gout Flares
Description: Count of gout flares
Time Frame: Day 90
Population: Due to study termination and small sample size, no analysis was performed
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year post randomization
Description: Clinicaltrials.gov definitions used.
Arm/Group | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 2/2 | 2/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) (N=2) | Placebo (N=2)
Esophageal Obstruction/Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Admitted for Esophageal obstruction, later diagnosed with esophageal cancer
PEG Placement (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abdominal Pain/Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute Chronic Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) — Fluid overload
Sub Therapeutic INR (Cardiac disorders) | 1 (1) | 0 (0)
Acute on Chronic Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
MRSA Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) (N=2) | Placebo (N=2)
Non-Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sub-Therapeutic INR (Cardiac disorders) | 2 (2) | 1 (1)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LAVD Alarm Issue (Cardiac disorders) | 0 (0) | 1 (2)
PICC Line Replacement (Infections and infestations) | 0 (0) | 1 (1)
Back/Shoulder/Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to lack of funding and COVID-19, the study was terminated early after 4 patients were recruited. This number is too small to perform any analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT03925324/Prot_SAP_000.pdf